CLINICAL TRIAL: NCT04864392
Title: A 5-year, Randomized, Double-blind, Placebo-controlled, Multi-center Study Assessing the Efficacy, Safety, and Tolerability of Intra-articular Regimens of LNA043 Versus Placebo in Patients With Symptomatic Knee Osteoarthritis
Brief Title: Study of Efficacy, Safety, and Tolerability of LNA043 in Patients With Knee Osteoarthritis
Acronym: ONWARDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study early terminated due to lack of effect (did not meet primary/key secondary endpoints). This decision was not linked to safety concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNA043A12202; 2020-004897-22 (EudraCT Number); 2023-509937-37-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2021-02-26; First posted 2021-04-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis
Keywords: LNA043; knee; arthritis; OA; knees
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LNA043 Dosing Regimen A (Experimental): LNA043 injection to the knee with dosing regimen A
  Interventions: Drug: LNA043 Dosing Regimen A
- LNA043 Dosing Regimen B (Experimental): LNA04 injection to the knee with dosing regimen B
  Interventions: Drug: LNA043 Dosing Regimen B
- LNA043 Dosing Regimen C (Experimental): LNA043 injection to the knee with dosing regimen C
  Interventions: Drug: LNA043 Dosing Regimen C
- LNA043 Dosing Regimen D (Experimental): LNA043 injection to the knee with dosing regimen D
  Interventions: Drug: LNA043 Dosing Regimen D
- Placebo (Placebo Comparator): Injection to the knee
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LNA043 Dosing Regimen A — Injection to the knee
  Other Names: LNA043
  Arms: LNA043 Dosing Regimen A
Drug: LNA043 Dosing Regimen B — Injection to the knee
  Other Names: LNA043
  Arms: LNA043 Dosing Regimen B
Drug: LNA043 Dosing Regimen C — Injection to the knee
  Other Names: LNA043
  Arms: LNA043 Dosing Regimen C
Drug: LNA043 Dosing Regimen D — Injection to the knee
  Other Names: LNA043
  Arms: LNA043 Dosing Regimen D
Drug: Placebo — Injection to the knee
  Arms: Placebo

SUMMARY:
The study will determine the optimal dosing regimen of LNA043 in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This study is a 2-period, multicenter, randomized, parallel-group, double-blind, placebo-controlled study consisting of a 2-year Core period, followed by a 3 year extension period. The primary objective of this study is to assess the efficacy of LNA043 compared to placebo at Week 104 as measured by the mean change from baseline in cartilage thickness using qMRI of the target knee

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 40 and 75 years of age
* Body mass index (BMI) < 40 kg/m2
* Diagnosis of primary tibiofemoral knee OA by standard American College of Rheumatology clinical and radiographic criteria
* and other criteria as specified by the protocol

Exclusion Criteria:

* Participants with radiographic knee OA K-L grade = 4 on the non-target knee
* Arthroscopy of the target knee within the 6 months prior to Screening
* Hemoglobin < 8.5 g/dL (85 g/L) or platelet count < 100,000/μL
* and other criteria as specified by the protocol

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the cartilage thickness of the medial compartment of the knee as assessed by imaging. | Week 0 to Week 104
  To evaluate cartilage thickness changes

SECONDARY OUTCOMES:
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index pain scale. The scale (5 questions) ranges from 0 to 50. Higher score indicates a worse outcome. | Week 0 to Week 104
  To evaluate changes from baseline in OA pain
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index function scale. The scale (17 questions) ranges from 0 to 170. Higher scores indicates a worse outcome. | Week 0 to Week 104
  To evaluate changes from baseline in physical function
Change from baseline in the cartilage thickness of the knee as assessed by imaging. | Week 0 to Week 104
  To evaluate changes from baseline the cartilage structure
Change from baseline in the Osteoarthritis Research Society International physical performance-based assessment of 40-meter (4×10m) fast-paced walk test | Week 0 to Week 104
  To evaluate changes from baseline in physical function
Change from baseline in the Osteoarthritis Research Society International physical performance-based assessments 30-second chair stand test | Week 0 to Week 104
  To evaluate changes from baseline in physical function
Change from baseline in the Osteoarthritis Research Society International physical performance-based assessment of 6-minute walking test | Weeek 0 to Week 104
  To evaluate changes from baseline in physical function
Proportion of participants demonstrating structural progression | Week 0 to Week 104
  To evaluate structural progression
Assessing percentage of participants with adverse events and serious adverse events | Week 0 to Week 104
  To evaluate safety and tolerability of the various LNA043 regimens

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (76):
- United States (23):
  - Elite Clinical Studies, Phoenix, Arizona
  - Tucson Orthopedic Institute PC, Tucson, Arizona
  - Sharps Hospital Grossmont, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - Long Beach Clinical Trials, Long Beach, California
  - Artemis Institute Clinical Research, Riverside, California
  - Northern California Research, Sacramento, California
  - Arthemis Clinical Research, San Diego, California
  - Stamford Therapeutics Consortium LLC, Stamford, Connecticut
  - Sensible Healthcare, Ocoee, Florida
  - Clinical Research of West Florida Inc, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Chicago Clinical Research Inst, Chicago, Illinois
  - Tandem clinical research, Marrero, Louisiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Center For Pharmaceutical Research, Kansas City, Missouri
  - Drug Trials America, Hartsdale, New York
  - AMR Knoxville, Knoxville, Tennessee
  - Metroplex Clinical Research, Dallas, Texas
  - Pioneer Research Solutions, Sugar Land, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Annapolis Rheumatology LLC, Fairfax, Virginia
  - Virginia Ispine Physicians PC, Richmond, Virginia
- Argentina (3):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, San Miguel de Tucumán
- Australia (8):
  - Novartis Investigative Site, Broadmeadow, New South Wales
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Woodville South, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern East, Victoria
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, St Leonards
  - Novartis Investigative Site, Waikanae Beach
- Canada (2):
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- China (2):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Bengbu
- Czechia (6):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Brno-Zidonice, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Denmark (3):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Gandrup
  - Novartis Investigative Site, Vejle
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- India (4):
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Pune
- Japan (5):
  - Novartis Investigative Site, Shinagawa, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Suginami, Tokyo
  - Novartis Investigative Site, Chuoh-ku
  - Novartis Investigative Site, Osaka
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Ciudad de
- Poland (4):
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Spain (6):
  - Novartis Investigative Site, Santiago de Compostela, A Coruna
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
- Taiwan (2):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Tainan
- United Kingdom (3):
  - Novartis Investigative Site, Barnet
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gerwin N, Scotti C, Halleux C, Fornaro M, Elliott J, Zhang Y, Johnson K, Shi J, Walter S, Li Y, Jacobi C, Laplanche N, Belaud M, Paul J, Glowacki G, Peters T, Wharton KA Jr, Vostiar I, Polus F, Kramer I, Guth S, Seroutou A, Choudhury S, Laurent D, Gimbel J, Goldhahn J, Schieker M, Brachat S, Roubenoff R, Kneissel M. Angiopoietin-like 3-derivative LNA043 for cartilage regeneration in osteoarthritis: a randomized phase 1 trial. Nat Med. 2022 Dec;28(12):2633-2645. doi: 10.1038/s41591-022-02059-9. Epub 2022 Dec 1. PMID 36456835